CLINICAL TRIAL: NCT04319146
Title: Pilot Feasibility Study of Robot-assisted Radical Prostatectomy Performed on Outpatient in Patients With Localized Prostate Cancer
Brief Title: Study of Robot-assisted Radical Prostatectomy Performed on Outpatient in Patients With Localized Prostate Cancer
Acronym: AMBUPRO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-AOIP-03
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label, monocentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- robot-assisted radical prostatectomy (Other): patient with a prostate cancer will be operated with a robot-assisted method. They will be supported on an outpatient basis
  Interventions: Procedure: robot-assisted radical prostatectomy

INTERVENTIONS:
Procedure: robot-assisted radical prostatectomy — robot-assisted radical prostatectomy as first-line treatment

SUMMARY:
The promoter propose a pilot study evaluating the feasability of robot-assisted radical prostatectomy on outpatient in patients with localized prostate cancer. This study will enrole a total of 20 patients over one center, followed for 1 month. The total study duration will be 15 months, including statistical analysis and publication.

DETAILED DESCRIPTION:
The promoter propose to carry out a monocentric biomedical cohort study, interventional, falling within the scope of the law of the public health code of 9 August 2004, for a total duration of 15 months including statistical analysis and publication. This analysis will involve a total of 20 patients, followed for 1 month during which the study criteria will be evaluated.

The patients concerned are men over 18 years of age (with a favourable onco-geriatric opinion if >70 years) with localised prostate cancer who are candidates for treatment by radical prostatectomy as first-line treatment. Patients must have a BMI of less than 35 kg/m², an ASA score of less than 3 and signed consent. Patients with a history of major abdominal surgery or sleep apnea syndrome will not be eligible.

The success rate of robot-assisted radical prostatectomy on an outpatient basis is defined by the absence of admission to a conventional inpatient unit within the first 24 hours after the procedure; the admission criterion being a Chung score of >9 (street-readiness score) or a complication during the procedure that does not allow the patient to be discharged.

Concerning post-operative follow-up, on D+1, readmissions and complications will be sought by the RAAC coordination nurse. The patient will be seen again at 1 month, during which time possible consultations and/or readmissions for events related to the operation will be sought. Urinary incontinence will be investigated by completing the ICIQ continence questionnaire and early oncological findings (PAS and histology of the surgical specimen) will be evaluated. Patient satisfaction with ambulatory surgery will be assessed using the SSQ8 questionnaire collected at this visit.

Investigators are selected on the basis of their surgical experience for this technique and must have performed a minimum of 20 personal procedures.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Older than 18 years old, if> 70 years old, then patient having had a favorable onco-geriatric consultation (Balducci 2 and life expectancy> 10 years)
* Patient with localized prostate cancer applying for radical prostatectomy treatment
* Patient accepting outpatient surgery
* Radical prostatectomy performed as first-line treatment
* BMI <35
* ASA score <3
* Accompanying person available (taxi authorized) to ensure return home
* Have quick access to a telephone line
* Patient who signed their informed consent
* Patient covered by social security or other health insurance

Exclusion Criteria:

* History of major abdominal surgery
* History of pelvic radiotherapy
* History of major urogenital malformation
* Sleep apnea syndrome
* Taking the following drugs within 48 hours (Plavix®, anti-vitamin K / curative LMWH)
* Contraindication to ambulatory medical care
* Inability to understand and sign the informed consent and to complete the self-questionnaires
* Vulnerable people

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Absence of conventional hospitalization after robot-assisted radical prostatectomy | 24 hours following the intervention

SECONDARY OUTCOMES:
Outpatient failure defined by a Chung score of less than 9 who cannot be discharged or admitted to a conventional hospitalization. | 24 hours following the intervention
Mesure of the operation duration will be estimated in minutes and will be recorded with a stopwatch in the operating room | The day of surgery
  Start = time of the incision, End = skin closure
The complication rate is determined by the number of patients who had one or more complications in the first month following the operation. Complications will be graded according to the Clavien Dindo classification. | within the month after surgery
The consultation rate in a doctor's office is set by the number of patients who consulted a general practitioner in the first month after the operation, declared by the patient during the control visite (at 1 month) | one month after surgery
•Any form of admission for urological reasons judged by the investigator in relation to robot-assisted radical prostatectomy within one month after the operation is considered as early unscheduled re-hospitalisation. | one month after surgery
Urinary incontinence is assessed by the ICIQ questionnaire at Month 1. | one month after surgery
  ICIQ is the incontinence international questionnaire used to evaluate the frequence, quantity and the interference of urine leakage. There are 3 questions and the sum of their answers gives the ICIQ score (between 0 and 21)
Patient satisfaction is assessed using the SSQ8 at Month 1. | one month after surgery
  SS8 is the Surgical Satisfaction questionnaire. There are 8 questions and the possible answers are Very satisfied, Sitisfied, Neutral, Unsatisfied, Very unsatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE Pasteur 2, Nice, CHU de Nice, France

IPD SHARING:
Plan to Share IPD: No
no plan description is necessary